CLINICAL TRIAL: NCT04475575
Title: Can the Electronic Nose Smell COVID-19 Antibodies? A Proof-of-principle Study
Brief Title: Can the Electronic Nose Smell COVID-19 Antibodies?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Nicole Bouvy, Prof. Dr. Nicole D. Bouvy, Maastricht University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: eNoseCOVIDantibodies
Record Dates: First submitted 2020-07-15; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: SARS-CoV Infection; Covid19
Keywords: Electronic nose; Volatile organic compounds; Diagnosis; Serology; Antibodies
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19; Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 suspected (Other): Participants where included if an oropharyngeal and nasopharyngeal swab was collected for RT-PCR and serology testing had been performed, or if participants have had a confirmed COVID-19 diagnosis in the previous days or weeks with an indication for re-testing via PCR and serology testing at the moment of inclusion
  Interventions: Device: Aeonose

INTERVENTIONS:
Device: Aeonose — All participants breathed through the Aeonose for five minutes. This device contains metal-oxide sensors that change in conductivity upon reaction with VOCs in exhaled breath. These conductivity changes are input data for machine-learning and used for pattern recognition. A nose clip was placed on the nose of each participant to avoid entry of non-filtered air in the device. Before measuring, the Aeonose was flushed with room air, guided through a carbon filter as well. During each measurement, a video was displayed to distract the participant and to reduce the chance of hyperventilation. Failed breath tests were excluded from analysis; the reason for failure was documented. Four similar Aeonose devices were used for breath analysis. A full-measurement procedure required sixteen minutes.

SUMMARY:
Corona Virus Disease (COVID-19), spread worldwide and has become an emergency of major international concern. In March 2020, the WHO declared the COVID-19 outbreak a global pandemic. Accurate and fast diagnosis is crucial in managing the pandemic. Current diagnostic approaches raise several difficulties: they are time-consuming, expensive, invasive, and most important lacking high sensitivity. The gold standard diagnostic test for COVID-19, reverse transcription polymerase chain reaction (RT-PCR), is highly dependent on adequate deep sampling of the swab in the naso- and oropharynx. A new diagnostic test that can correctly and rapidly identify infected patients and asymptomatic carriers is urgently required to prevent further virus transmission and thus reduce mortality rates.

Aim: This proof-of-principle study aims to investigate if an electronic nose (Aeonose) can distinguish individuals with antibodies from individuals without antibodies against COVID-19 based on analysis of volatile organic compounds (VOCs).

Methods: between April and July 2020, persons undergoing RT-PCR and a serology test for COVID-19 were recruited at Maastricht UMC+ for breath analysis. All participants had to breathe through the Aeonose for five consecutive minutes. The VOC pattern in their exhaled breath was then linked to the matching RT-PCR and serological test results.

ELIGIBILITY:
Inclusion Criteria:

* Participants of whom an oropharyngeal and nasopharyngeal swab was collected for RT-PCR and on whom serology testing for the detection of antibodies was performed.

Exclusion Criteria:

* Participants who where experiencing dyspnea or needed supplemental oxygen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
COVID-19 antibodies vs COVID-19 negative | 3 months
  Ability of the electronic nose (Aeonose) to distinguish individuals with antibodies from individuals without antibodies against COVID-19 based on analysis of volatile organic compounds (VOCs).

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] de Lacy Costello B, Amann A, Al-Kateb H, Flynn C, Filipiak W, Khalid T, Osborne D, Ratcliffe NM. A review of the volatiles from the healthy human body. J Breath Res. 2014 Mar;8(1):014001. doi: 10.1088/1752-7155/8/1/014001. Epub 2014 Jan 13. PMID 24421258
- [Background] Xiang F, Wang X, He X, Peng Z, Yang B, Zhang J, Zhou Q, Ye H, Ma Y, Li H, Wei X, Cai P, Ma WL. Antibody Detection and Dynamic Characteristics in Patients With Coronavirus Disease 2019. Clin Infect Dis. 2020 Nov 5;71(8):1930-1934. doi: 10.1093/cid/ciaa461. PMID 32306047
- [Background] Schuermans VNE, Li Z, Jongen ACHM, Wu Z, Shi J, Ji J, Bouvy ND. Pilot Study: Detection of Gastric Cancer From Exhaled Air Analyzed With an Electronic Nose in Chinese Patients. Surg Innov. 2018 Oct;25(5):429-434. doi: 10.1177/1553350618781267. Epub 2018 Jun 18. PMID 29909757
- [Background] Bikov A, Lazar Z, Horvath I. Established methodological issues in electronic nose research: how far are we from using these instruments in clinical settings of breath analysis? J Breath Res. 2015 Jun 9;9(3):034001. doi: 10.1088/1752-7155/9/3/034001. PMID 26056127
- [Background] Bijland LR, Bomers MK, Smulders YM. Smelling the diagnosis: a review on the use of scent in diagnosing disease. Neth J Med. 2013 Jul-Aug;71(6):300-7. PMID 23956311
- [Background] van Geffen WH, Bruins M, Kerstjens HA. Diagnosing viral and bacterial respiratory infections in acute COPD exacerbations by an electronic nose: a pilot study. J Breath Res. 2016 Jun 16;10(3):036001. doi: 10.1088/1752-7155/10/3/036001. PMID 27310311